CLINICAL TRIAL: NCT04084002
Title: Evaluation of Physical Activity and Related Factors in a Sample of Turkish Patients With Stroke
Brief Title: Physical Activity and Related Factors in a Sample of Turkish Patients With Stroke
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Marmara University (Other)
Responsible Party: Sponsor
Other Study IDs: 17.12.2018-242
Record Dates: First submitted 2019-09-06; First posted 2019-09-10 (Actual); Last update posted 2019-09-17 (Actual); Status verified 2019-09

CONDITIONS: Stroke
Keywords: stroke; physical activity
MeSH Terms: conditions — Stroke; Motor Activity | interventions — Exercise

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with subacute chronic stroke: Patients with subacute chronic stroke
  Interventions: Other: physical activity measurement
- Control group: Healthy control group age and sex matched
  Interventions: Other: physical activity measurement

INTERVENTIONS:
Other: physical activity measurement — Physical activity will be measured via accelerometer and self reported questionnaire (Physical activity scale for elderly)

SUMMARY:
The aim of this study was to investigate the relationships between physical activity level and demographic factors, motor function, cognitive function, functional status, balance and quality of life in patients with chronic stroke and to compare physical activity levels with healthy individuals in the same population.

DETAILED DESCRIPTION:
The aim of this study was to investigate the relationships between physical activity level and demographic factors, motor function, cognitive function, functional status, balance and quality of life in patients with chronic stroke and to compare physical activity levels with healthy individuals in the same population. It is a fact that the physical activity levels of individuals decrease significantly after stroke. However, there is no study examining to what extent the physical activity is affected and the factors related to the decrease in the level of physical activity. The primary aim of stroke rehabilitation is to recognize and prevent complications, to minimize disturbances, to maximize functions. Secondary objectives; to prevent stroke recurrence. Physical activity has been shown to reduce the risk of stroke, stroke severity and other consequences. The risk of a reduction in physical capacity occurs over time and it is assumed that normal physical activity can prevent recurrent stroke. Therefore, it is necessary to continuously assess physical activity levels after stroke. In order to increase physical activity levels, it is important to identify people with low levels of physical activity and to understand the factors that may be associated. Therefore, in this study, we aimed to provide a comprehensive analysis by including most of the factors that may be related to physical activity in patients with stroke. In this study, unlike previous studies on physical activity in stroke, the relationships between physical activity and factors such as motor function, quality of life and cognitive skills as well as balance measurements and walking speed parameters which will be obtained from computerised posturography will be examined. In previous studies Physical Activity Scale for Elderly (PASE) questionnaire or the accelerometer device are used for the measurement of physical activity level. In this study, both of these tools will be used and the correlation between these two assessment tools will be demonstrated. In this study, patients with stroke will be evaluated by using PASE scale and accelerometer results (accelerometer will be held from Monday to Friday) for physical activity and Mini Mental test for cognitive function, Fugl Meyer Scale for motor function, Berg Balance Test and computerized posturography analysis for balance, Barthel Index for daily activities, Stroke Impact Scale for quality of life, Brunnstrom stage for motor recovery status. Each of the tests lasts about 5-10 minutes. Healthy control group will also be assessed via accelerometer and PASE questionnaire for physical activity and computerized posturography for balance.

With this study, physical activity which is protective for recurrent stroke, will be evaluated comprehensively and factors associated with physical activity will be revealed. Thus, in order to increase the physical activity, it will be concluded which factor should be treated or evaluated, and these results will be very helpful for further studies.

ELIGIBILITY:
Inclusion Criteria:

Patient group

1. Patients with first ever, unilateral stroke
2. Patients with stroke who can walk independently or with an assistive device
3. Being at between the ages of 40-80 Control group

1. Being at between the ages of 40-80 and having not previously diagnosed with any neurologic disease

Exclusion Criteria:

Patient group

1. Having uncontrolled hypertension, cardiopulmonary disease
2. Presence of neglect, dementia, apraxia
3. Mini mental scale >24 or being able to complete study outcomes

Ages: 40 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with stroke and their age and sex matched controls
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-09-16 (Actual); Primary Completion 2019-11-15 (Estimated); Study Completion 2019-11-16 (Estimated)

PRIMARY OUTCOMES:
ACtotal | Day 0
  Total activity count (AC) obtained from accelerometer
EEtotal | Day 0
  Total energy expenditure (EE) obtained from accelerometer
PASE | Day 0
  Physical Activity Score for Elderly (PASE)

SECONDARY OUTCOMES:
AC moderate | Day 0
  activity counts derived from accelerometer during moderate physical activity
EE moderate | Day 0
  energy expenditure obtained from accelerometer during moderate physical activity
AC light | Day 0
  activity counts derived from accelerometer during light physical activity
EE light | Day 0
  energy expenditure obtained from accelerometer during light physical activity
AC vigorous | Day 0
  activity counts derived from accelerometer during vigorous physical activity
EE vigorous | Day 0
  energy expenditure obtained from accelerometer during vigorous physical activity
AC sedentary | Day 0
  activity counts derived from accelerometer during sedentary physical activity
EE sedentary | Day 0
  energy expenditure obtained from accelerometer during sedentary physical activity
step count | Day 0
  total step count obtained from accelerometer
Stroke Impact Scale | Day 0
  Stroke Impact Scale
Berg Balance Score | Day 0
  Berg Balance Score
Barthel Index for Activities of Daily Living | Day 0
  Barthel Index for Activities of Daily Living
FMA-UE | Day 0
  The Fugl-Meyer Assessment for upper extremity
FMA-LE | Day 0
  The Fugl-Meyer Assessment for lower extremity
FMA-total | Day 0
  The Fugl-Meyer Assessment total score
Brunnstrom stage for proximal upper extremity | Day 0
  Brunnstrom stage for proximal upper extremity
Brunnstrom stage for distal upper extremity | Day 0
  Brunnstrom stage for distal upper extremity
Brunnstrom stage for lower extremity | Day 0
  Brunnstrom stage for lower extremity
FAS stage | Day 0
  Functional Ambulation Scale (FAS) stage
Mini Mental Test | Day 0
  Mini Mental Test
stroke duration | Day 0
  stroke duration
WA step width | Day 0
  Walk Across step width obtained from Neurocom forceplate
WA step length | Day 0
  Walk Across step width obtained from Neurocom forceplate
WA walking speed | Day 0
  Walk Across walking speed obtained from Neurocom forceplate
Modified Clinical Test of Sensory Interaction on Balance | Day 0
  Modified Clinical Test of Sensory Interaction on Balance obtained from Neurocom forceplate
LOS RT | Day 0
  Limits of Stability reaction time obtained from Neurocom forceplate
LOS VL | Day 0
  Limits of Stability movement velocity obtained from Neurocom forceplate
LOS EPE | Day 0
  Limits of Stability endpoint excursion obtained from Neurocom forceplate
LOS MXE | Day 0
  Limits of Stability maximum excursion obtained from Neurocom forceplate
LOS DCL | Day 0
  Limits of Stability directional control obtained from Neurocom forceplate

CONTACTS AND LOCATIONS:
Overall Officials: Evrim Karadag Saygi, Prof, Study Chair — Marmara University
Locations (1):
- Marmara University School of Medicine, Pendik Research and Education Hospital, Department of Physical Medicine and Rehabilitation, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Result] Danielsson A, Meirelles C, Willen C, Sunnerhagen KS. Physical activity in community-dwelling stroke survivors and a healthy population is not explained by motor function only. PM R. 2014 Feb;6(2):139-45. doi: 10.1016/j.pmrj.2013.08.593. Epub 2013 Aug 23. PMID 23978463
- [Result] Lacroix J, Daviet JC, Borel B, Kammoun B, Salle JY, Mandigout S. Physical Activity Level Among Stroke Patients Hospitalized in a Rehabilitation Unit. PM R. 2016 Feb;8(2):97-104. doi: 10.1016/j.pmrj.2015.06.011. Epub 2015 Jun 21. PMID 26107540